CLINICAL TRIAL: NCT05631171
Title: COVIDAI: Feasibility Study of Adhera® Fatigue Digital Program for Patients With Long COVID-related Fatigue
Brief Title: Feasibility Study of Adhera® Fatigue Digital Program for Patients With Long COVID-related Fatigue
Acronym: COVIDAI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adhera Health, Inc. (Industry)
Collaborators: Institut Català de la Salut (Other); Andaluz Health Service (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FAT-22-002
Record Dates: First submitted 2022-11-18; First posted 2022-11-30 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-01

CONDITIONS: Post-Acute COVID19 Syndrome; Fatigue
Keywords: Long COVID; digital health; fatigue; emotional health; behavioral intervention; mental wellbeing
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Fatigue; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Experimental intervention arm in parallel to control arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Solution group (Experimental): The study sample will consist of 60 patients, 30 of whom will be randomly assigned to a control group and 30 to the experimental group. Validated questionnaires will be administered to the participants of both groups, at the beginning of the study, at 1 month and 3 months by Microsoft Forms. In addition, the experimental group will be given a smartwatch to each person which will collect real-time data on activity, training and sleep in a completely anonymous way. Also, through a mobile application, the patient of the experimental group will answer questionnaires about health status perception. The application has also been trained to provide educational content and motivational messages to support the patient's self-management. The data provided by patients in both groups of the study will be coded, in order to maintain the confidentiality of the individual.
  Interventions: Behavioral: Adhera® Fatigue Digital Program
- Control group (No Intervention): The study sample will consist of 60 patients, 30 of whom will be randomly assigned to a control group and 30 to the experimental group. Validated questionnaires will be administered to the participants of both groups, at the beginning of the study, at 1 month and 3 months by Microsoft Forms.

INTERVENTIONS:
Behavioral: Adhera® Fatigue Digital Program — Adhera® Fatigue Digital Program, that includes an application and a smartwatch, is a digital health solution based on emotional and behavioral change techniques. Patient adaptative self-management content (e.g. psycho-educational content, activities for mental wellbeing, personalized motivational messages), and the personalization is based on Adhera® Health Recommender System.
  Wearable devices and the mobile app will be used to collect real-time data for 3 months to detect biometric and psychometric (patient-reported outcomes) information.
  Arms: Solution group

SUMMARY:
Adhera® Fatigue Digital Program (or AFDP) is a digital health program based on behavioral and emotional change techniques that provides personalized physical and emotional self-management support for patients with long COVID-related fatigue.

The digital health solution is designed to be used for 3 months, and includes a mobile application and a smartwatch. This is a clinical study, with 30 participants in the experimental intervention group and 30 in the control group, that will be carried out at the Jordi Gol Primary Care Research Institute (IDIAPJGol) - Institut Català de la Salut and Distrito sanitario Aljarafe-Sevilla Norte (DASN) - Servicio Andaluz de Salud, in Spain. The investigators will focus on evaluating the feasibility of the program in supporting fatigue and also physical and emotional self-management and, consequently, in improving the patients' well-being and quality of life.

DETAILED DESCRIPTION:
The COVIDAI study will collect data on symptomatology and emotional well-being in a population of patients with fatigue related to a diagnosis of long COVID for 3 months using or not using the Adhera® Fatigue Digital Program (30 participants in the experimental intervention group and 30 in the control group). The aim of the study is to evaluate the feasibility of the program in supporting physical and emotional self-management in long COVID patients with fatigue and, consequently, in improving the patients' quality of life.

Personalized digital health solutions for both physiological and psychological long COVID-related symptoms would allow an optimization of the cost-effectiveness model for the management of long COVID patients. Similarly, the early detection of complications associated to long COVID on patients from vulnerable groups would improve the care timeline and the patient's prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Individuals over 18 years of age.
* With long COVID, according to the World Health Organization (WHO) consensus definition
* Having a history of fatigue symptoms
* Obtain a score between 4 and 10 on the question "By how much do you rate your fatigue level from 0 to 10 in the last 7 days?", where 0 is no fatigue and 10 is the worst fatigue imaginable
* Have an Android or iOS smartphone compatible with the intervention program.
* Agree to participate in the study and sign the informed consent form
* Willingness and availability to comply with all study guidelines and procedures

Exclusion Criteria:

* Hospital admission during the period of study participation.
* Participation in another study with pharmacological treatment
* Patients who are not technologically literate or unable to use the mobile application.
* Known severe psychiatric illness or presence of relevant cognitive impairment, at the discretion of the recruiting physician
* With mobility restrictions that limit the patient's ability to perform mild physical activity
* Being pregnant
* Patients who do not understand or speak Catalan or Spanish.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2022-12-13 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Health-related quality of life | baseline
  measured using the 5-level EQ-5D (EQ-5D-5L) questionnaire from Herdman et al., 2011. Health state index scores generally range from less than 0 (where 0 is the value of a health state equivalent to dead; negative values representing values as worse than dead) to 1 (the value of full health), with higher scores indicating higher health utility.
Health-related quality of life | month 1
  measured using the 5-level EQ-5D (EQ-5D-5L) questionnaire from Herdman et al., 2011. Health state index scores generally range from less than 0 (where 0 is the value of a health state equivalent to dead; negative values representing values as worse than dead) to 1 (the value of full health), with higher scores indicating higher health utility.
Health-related quality of life | month 3
  measured using the 5-level EQ-5D (EQ-5D-5L) questionnaire from Herdman et al., 2011. Health state index scores generally range from less than 0 (where 0 is the value of a health state equivalent to dead; negative values representing values as worse than dead) to 1 (the value of full health), with higher scores indicating higher health utility.
Fatigue | baseline
  Perceived mental and physical fatigue will be assessed via the Fatigue Assessment Scale (FAS), from De Vries et al., 2004. The total score ranges from 10 to 50, with a higher score indicating more severe fatigue.
Fatigue | month 1
  Perceived mental and physical fatigue will be assessed via the Fatigue Assessment Scale (FAS), from De Vries et al., 2004. The total score ranges from 10 to 50, with a higher score indicating more severe fatigue.
Fatigue | month 3
  Perceived mental and physical fatigue will be assessed via the Fatigue Assessment Scale (FAS), from De Vries et al., 2004. The total score ranges from 10 to 50, with a higher score indicating more severe fatigue.
Emotional wellness | baseline
  measured using the Depression Anxiety Stress Scale (DASS-21) from Lovibond, 1995. Scoring ranges from 0 to more than 34, with the lowest numbers being the normal ones and the highest representing extremely severe depression, anxiety and stress.
Emotional wellness | month 1
  measured using the Depression Anxiety Stress Scale (DASS-21) from Lovibond, 1995. Scoring ranges from 0 to more than 34, with the lowest numbers being the normal ones and the highest representing extremely severe depression, anxiety and stress.
Emotional wellness | month 3
  measured using the Depression Anxiety Stress Scale (DASS-21) from Lovibond, 1995. Scoring ranges from 0 to more than 34, with the lowest numbers being the normal ones and the highest representing extremely severe depression, anxiety and stress.

SECONDARY OUTCOMES:
Behavioral outcome: Usability | month 1
  Digital health solution usability and acceptance assessed with the System Usability Scale (SUS) questionnaire from Bangor et al., 2008. SUS can range between score 0 and 100, with higher values representing higher usability.
Behavioral outcome: Usability | month 3
  Digital health solution usability and acceptance assessed with the System Usability Scale (SUS) questionnaire from Bangor et al., 2008. SUS can range between score 0 and 100, with higher values representing higher usability.
Fatigue-related symptomatology | month 1
  questions regarding perceived anxiety, depression, stress, sleep disorders or emotional status.
Fatigue-related symptomatology | month 3
  questions regarding perceived anxiety, depression, stress, sleep disorders or emotional status.
Mood | baseline
  measured using the Positive and Negative Affect Schedule (PANAS) from Watson et al., 1988. Positive Affect Score can range from 10 - 50, with higher scores representing higher levels of positive affect. Negative Affect Score can range from 10 - 50, with lower scores representing lower levels of negative affect.
Mood | month 1
  measured using the Positive and Negative Affect Schedule (PANAS) from Watson et al., 1988. Positive Affect Score can range from 10 - 50, with higher scores representing higher levels of positive affect. Negative Affect Score can range from 10 - 50, with lower scores representing lower levels of negative affect.
Mood | month 3
  measured using the Positive and Negative Affect Schedule (PANAS) from Watson et al., 1988. Positive Affect Score can range from 10 - 50, with higher scores representing higher levels of positive affect. Negative Affect Score can range from 10 - 50, with lower scores representing lower levels of negative affect.
Social, psychological and emotional wellness | baseline
  Mental Health Continuum Short Form (MHC-SF) from Keyes et al., 2008. Items are summed, yielding a total score ranging from 0 to 70. Subscale scores range from 0 to 15 for the emotional (hedonic) well-being, from 0 to 25 for social well-being, and from 0 to 30 for psychological well-being. Flourishing mental health is defined by reporting ≥ 1 of 3 hedonic signs and ≥ 6 of 11 eudaimonic signs (social and psychological subscales combined) experienced "every day" or "5-6 times a week." Higher scores indicate greater levels of positive well-being.
Social, psychological and emotional wellness | month 1
  Mental Health Continuum Short Form (MHC-SF) from Keyes et al., 2008. Items are summed, yielding a total score ranging from 0 to 70. Subscale scores range from 0 to 15 for the emotional (hedonic) well-being, from 0 to 25 for social well-being, and from 0 to 30 for psychological well-being. Flourishing mental health is defined by reporting ≥ 1 of 3 hedonic signs and ≥ 6 of 11 eudaimonic signs (social and psychological subscales combined) experienced "every day" or "5-6 times a week." Higher scores indicate greater levels of positive well-being.
Social, psychological and emotional wellness | month 3
  Mental Health Continuum Short Form (MHC-SF) from Keyes et al., 2008. Items are summed, yielding a total score ranging from 0 to 70. Subscale scores range from 0 to 15 for the emotional (hedonic) well-being, from 0 to 25 for social well-being, and from 0 to 30 for psychological well-being. Flourishing mental health is defined by reporting ≥ 1 of 3 hedonic signs and ≥ 6 of 11 eudaimonic signs (social and psychological subscales combined) experienced "every day" or "5-6 times a week." Higher scores indicate greater levels of positive well-being.
Self-efficacy | baseline
  Self-Efficacy Scale (GSE) from Schwartzer & Jerusalem 1995. The total score ranges between 10 and 40, with a higher score indicating more self-efficacy.
Self-efficacy | month 1
  Self-Efficacy Scale (GSE) from Schwartzer & Jerusalem 1995. The total score ranges between 10 and 40, with a higher score indicating more self-efficacy.
Self-efficacy | month 3
  Self-Efficacy Scale (GSE) from Schwartzer & Jerusalem 1995. The total score ranges between 10 and 40, with a higher score indicating more self-efficacy.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Gerencia Territorial de la Catalunya Central - Institut Catala de la Salut, Sant Fruitós de Bages, Barcelona
  - Servicio Andaluz de Salud - Distrito Sanitario Aljarafe-Sevilla Norte, Seville

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Withings Scanwatch wearable — https://www.withings.com/de/en/scanwatch